CLINICAL TRIAL: NCT03885284
Title: Phase I Study of Proton Therapy in Adjuvant Pancreatic Cancer (Proton-PANC)
Brief Title: Study of Proton Therapy in Adjuvant Pancreatic Cancer
Acronym: Proton-PANC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1021
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2023-11

CONDITIONS: Resected Pancreatic Adenocarcinoma
Keywords: Pancreas; Radiation; mFOLFIRINOX
MeSH Terms: interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dose Level 1 (Experimental): mFOLFIRINOX + Proton beam radiation
  Radiation given on days 8-12 of cycle 6
  Interventions: Drug: mFOLFIRINOX; Radiation: Proton beam radiation
- Dose Level 2 (Experimental): mFOLFIRINOX + Proton beam radiation
  Radiation given on days 15-19 of cycle 6
  Interventions: Drug: mFOLFIRINOX; Radiation: Proton beam radiation

INTERVENTIONS:
Drug: mFOLFIRINOX — Chemotherapy will consist of mFOLFIRINOX in 14-day cycles x 12 as used in the PRODIGE 24 study:
  * Irinotecan 150 mg/m2 IV day 1
  * Oxaliplatin 85 mg/m2 IV day 1
  * Leucovorin 400 mg/m2 IV day 1
  * 5-fluorouracil 2,400 mg/m2 IV days 1-3 (no bolus)
  * Pegfilgrastim 6 mg SC on-body injector day 3 (optional, up to investigator's discretion, can alternatively do day 4 without on-body injector)
  * Suggested supportive care medications: fosaprepitant 150 mg IV day 1, dexamethasone 12 mg IV day 1, ondansetron 16 mg IV day 1, dexamethasone 4 mg PO q AM days 2-3, ondansetron 8 mg PO BID days 2-3.
Radiation: Proton beam radiation — Proton beam radiation will consist of 5 daily doses of 5 GyE total, ideally administered Monday through Friday but can be administered within 7 business days, between cycles 6 and 7

SUMMARY:
This trial aims to determine a safe schedule of short-course proton beam radiation therapy with adjuvant mFOLFIRINOX for patients with resected pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
The investigators hypothesize that resected pancreatic cancer patients will benefit from enhanced local control with the addition of radiation therapy to adjuvant FFX. The recently reported PRODIGE 24 study, demonstrated that 12 cycles of adjuvant FFX without radiation therapy significantly improved survival and time to metastatic failure rates as compared to GEM alone. Excessive distant failures rates using prior adjuvant systemic therapies, may have limited the impact of radiation therapy; therefore, improvements in systemic control can increase the benefit of local control.

In this study, the investigators utilize 5 fraction PRT, delivered over 1 week, during adjuvant FFX (between cycles 6 and 7) to minimize the interruptions in chemotherapy as well as to reduce the length of time from surgical resection to initiating adjuvant radiation therapy. Conventional radiation therapy is typically delivered over 5 weeks and is commonly given after the completion of adjuvant chemotherapy. Conventional radiation therapy cannot be given concurrently with FFX due to the synergistic toxicities. In contrast, PRT significantly reduces the exposure of normal tissues to the effects of radiation therapy and has been safely delivered using a 5 fraction schedule with chemotherapy, as previously discussed.

Chemotherapy will consist of mFOLFIRINOX in 14-day cycles x 12 as used in the PRODIGE 24 study:

* Irinotecan 150 mg/m2 IV day 1
* Oxaliplatin 85 mg/m2 IV day 1
* Leucovorin 400 mg/m2 IV day 1
* 5-fluorouracil 2,400 mg/m2 IV days 1-3 (no bolus)
* Pegfilgrastim 6 mg SC on-body injector day 3 (optional, up to investigator's discretion, can alternatively do day 4 without on-body injector)
* Suggested supportive care medications: fosaprepitant 150 mg IV day 1, dexamethasone 12 mg IV day 1, ondansetron 16 mg IV day 1, dexamethasone 4 mg PO q AM days 2-3, ondansetron 8 mg PO BID days 2-3.
* Dose adjustments will be permitted at the discretion of the treating oncologist based on patients' prior tolerability to FFX
* Proton radiation will consistent of 5 daily doses of 5 GyE total, ideally administered Monday through Friday but can be administered within 7 business days, between cycles 6 and 7

ELIGIBILITY:
Inclusion Criteria:

* Undergone pancreaticoduodenectomy with curative intent
* Pathologically-confirmed pancreatic adenocarcinoma of the pancreatic head (adenocarcinoma must be the predominant component of the histology)
* Completed 2 cycles of adjuvant chemotherapy composed of 5-fluorouracil, leucovorin, oxaliplatin, and irinotecan
* Complete resection (R0) or resection with microscopic positive magins (R1)
* Adequate healing post-operatively
* Bone marrow function: absolute neutrophil count (ANC) ≥ 1,500/mm3; Platelets ≥ 100 × 109/L; hemoglobin ≥ 9.0 g/dL. Patients may have a transfusion of red blood cells to meet the hemoglobin requirement.
* Renal function: serum creatinine ≤ 1.5 × upper normal limit of institution's normal range or creatinine clearance ≥ 30 mL/min for subjects with creatinine levels above institutional normal
* Hepatic function: AST and ALT ≤ 3.0 × the upper normal limit of institution's normal range. Total bilirubin ≤ 1.5 × the upper normal limit of institution's normal range.
* Partial Thromboplastin Time (PTT) must be ≤ 1.5 × upper normal limit of institution's normal range and INR (International Normalized Ratio) < 1.5. Subjects on anticoagulant (such as warfarin) will be permitted to enroll as long as the INR is in the acceptable therapeutic range as determined by the investigator.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0-1
* Prior neoadjuvant chemotherapy is alllowed
* Patients must have fully recovered from all effects of surgery. Patients must have had at least two weeks after minor surgery and four weeks after major surgery before starting therapy. Minor procedures requiring "Twilight" sedation such as endoscopies or mediport placement may only require a 24-hour waiting period, but this must be discussed with an investigator.
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to initiation of treatment and/or postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential
* Patient is capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent, approved by the Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures

Exclusion Criteria:

* Ampullary adenocarcinoma
* Women who are pregnant or breastfeeding
* Macroscopic positive margins (R2) or evidence of residual local or metastatic disease
* Resection not including pancreaticoduodenectomy
* Known allergy or intolerance to leucovorin, 5-fluorouracil, oxaliplatin, or irinotecan
* Prior radiation to the upper abdomen
* Inability to swallow pills or bowel obstruction
* Any invasive cancer in the previous 3 years requiring chemotherapy, radiation, or anticancer therapy following surgery
* Insurance unwilling to pre-authorize PRT, FFX, and (if necessary) pegfilgrastim
* Clinically significant liver disease (Patients with resolved hepatitis B infection are eligible if HBsAg testing is negative; Patients with resolved hepatitis C infection are eligible if viral RNA PCR is negative)
* Uncontrolled HIV infection (CD4 count must be at least 200 and viral load undectable on a stable antiretroviral regimen to be eligible for enrollment)
* Major surgery within 4 weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2023-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Weinberg, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: mFOLFIRINOX + Proton beam radiation
  Radiation given on days 8-12 of cycle 6
  mFOLFIRINOX: Chemotherapy will consist of mFOLFIRINOX in 14-day cycles x 12 as used in the PRODIGE 24 study:
  * Irinotecan 150 mg/m2 IV day 1
  * Oxaliplatin 85 mg/m2 IV day 1
  * Leucovorin 400 mg/m2 IV day 1
  * 5-fluorouracil 2,400 mg/m2 IV days 1-3 (no bolus)
  * Pegfilgrastim 6 mg SC on-body injector day 3 (optional, up to investigator's discretion, can alternatively do day 4 without on-body injector)
  * Suggested supportive care medications: fosaprepitant 150 mg IV day 1, dexamethasone 12 mg IV day 1, ondansetron 16 mg IV day 1, dexamethasone 4 mg PO q AM days 2-3, ondansetron 8 mg PO BID days 2-3.
  Proton beam radiation: Proton beam radiation will consist of 5 daily doses of 5 GyE total, ideally administered Monday through Friday but can be administered within 7 business days, between cycles 6 and 7
- Dose Level 2: mFOLFIRINOX + Proton beam radiation
  Radiation given on days 15-19 of cycle 6
  mFOLFIRINOX: Chemotherapy will consist of mFOLFIRINOX in 14-day cycles x 12 as used in the PRODIGE 24 study:
  * Irinotecan 150 mg/m2 IV day 1
  * Oxaliplatin 85 mg/m2 IV day 1
  * Leucovorin 400 mg/m2 IV day 1
  * 5-fluorouracil 2,400 mg/m2 IV days 1-3 (no bolus)
  * Pegfilgrastim 6 mg SC on-body injector day 3 (optional, up to investigator's discretion, can alternatively do day 4 without on-body injector)
  * Suggested supportive care medications: fosaprepitant 150 mg IV day 1, dexamethasone 12 mg IV day 1, ondansetron 16 mg IV day 1, dexamethasone 4 mg PO q AM days 2-3, ondansetron 8 mg PO BID days 2-3.
  Proton beam radiation: Proton beam radiation will consist of 5 daily doses of 5 GyE total, ideally administered Monday through Friday but can be administered within 7 business days, between cycles 6 and 7
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2
Started | 3 | 6
Completed | 2 | 2
Not Completed | 1 | 4
Not completed — Disease Progression | 1 | 3
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose Limiting Toxicites (DLTs)
Description: Recommended phase II dose and schedule (RP2D) of short-course PRT integrated within adjuvant mFOLFIRINOX will be based on number of Dose limiting toxicities.
Time Frame: 6 months
Measure: Number; unit: Dose limiting Toxicities
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 3 | 6
Dose limiting Toxicities | 0 | 1

2. Primary Outcome: Safety (Adverse Events) of Short-course PRT Integrated Within Adjuvant mFOLFIRINOX
Description: Dose Limiting Toxicities. Adverse Event data will be collected and presented as descriptive statistics using the CTCAE version 5.0
Time Frame: 6 months
Population: number of participants that had a dose limiting toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 3 | 6
Participants | 0 | 1

3. Primary Outcome: Feasibility (Rate of Successful Completion) of Short-course PRT Integrated Within Adjuvant mFOLFIRINOX
Description: Success rate defined as # of patients that completed proton beam planning, proton beam treatment, and completion of adjuvant therapy
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 3 | 6
Participants
  Completion PRT | 3 | 6
  completion of proton beam planning | 3 | 6
  completion of proton beam treatment | 3 | 6
  completion of adjuvant therapy | 2 | 2

4. Secondary Outcome: Recurrence-free Survival (RFS)
Description: Defined as time from surgery until evidence of disease recurrence.
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 3 | 6
months | 12 [4 to NA] — Upper Bound Not Reached due to insufficient number of participants with events | 12 [4 to NA] — Upper bound Not Reached due to insufficient number of participants with events

5. Secondary Outcome: Overall Survival (OS)
Description: Defined as time from surgery until death from any cause or last follow-up.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 3 | 6
Participants | 2 | 4

ADVERSE EVENTS:
Time Frame: AE and SAEs were collected from the time of study drug administration until 30 days following discontinuation of study drug administration (about 20 weeks). Deaths were assessed over 2 years.
Arm/Group | Dose Level 1 | Dose Level 2
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=6)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=6)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (3)
Pain (General disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (3)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 5 (6)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT03885284/Prot_SAP_000.pdf